CLINICAL TRIAL: NCT05229354
Title: Phase II Evaluation of the Safety and Protective Efficacy of a Single Dose of the Live Attenuated Tetravalent Dengue Vaccine TetraVax-DV TV005 to Protect Against Infection With Live, Recombinant DENV-2 (rDEN2∆30-7169) Attenuated Strain in a Dengue Endemic Population in South Asia
Brief Title: Dengue Controlled Human Infection Model in Dhaka, Bangladesh
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Beth Kirkpatrick (Other)
Collaborators: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Responsible Party: Sponsor-Investigator, Beth Kirkpatrick, MD, Professor of Medicine, University of Vermont
Organization: University of Vermont (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PR-19099
Record Dates: First submitted 2021-10-18; First posted 2022-02-08 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Dengue
MeSH Terms: conditions — Dengue

STUDY DESIGN:
Intervention Model Description: Eligible volunteers will be enrolled to receive TetraVax-DV TV005 or placebo (2:1) on an outpatient basis in one of three cohorts based on intended treatment with the attenuated virus strain timepoint (6, 12 or 24 months). The sequence of treatment assignments to either TV005 or placebo will be generated using block randomization. Randomization will occur sequentially at the time of study enrollment (vaccination) using a pre-generated list. All enrolled volunteers will be followed for 3 years post-vaccination for safety.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: While clinical staff, all investigators, and study volunteers will remain blinded until each cohort's respective unblinding timepoint, the PI will assign an unblinded statistician to analyze the safety data. This designee will provide safety data to study staff as a summary report with blinding maintained.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Intervention followed by challenge (Experimental): Participants receiving TV005 and then challenged with the rDEN2Δ30-7169 attenuated virus strain.
  Interventions: Biological: TV005; Biological: rDEN2Δ30-7169 attenuated virus strain
- Placebo followed by challenge (Experimental): Participants receiving placebo and then challenged with the rDEN2Δ30-7169 attenuated virus strain.
  Interventions: Biological: rDEN2Δ30-7169 attenuated virus strain

INTERVENTIONS:
Biological: TV005 — The TV005 admixture is comprised of four monovalent dengue vaccine candidates representing each of the four DENV serotypes: rDEN1Δ30, rDEN2/4Δ30(ME), rDEN3Δ30/31, and rDEN4Δ30.
  Arms: Intervention followed by challenge
Biological: rDEN2Δ30-7169 attenuated virus strain — based on a cDNA derived DENV-2 virus (strain Tonga/74) in which the 3´ UTR of DENV-2 contains a 30 (nt) deletion (nt 173 - 143) homologous to the ∆30 deletion in the 3´ UTR of rDEN4Δ30 (named Δ30 for consistency). A plasmid was constructed to encode the entire genome of DENV-2 Tonga/74. The cDNA of the 3´ UTR of DENV-2 Tonga/74 was then modified to introduce a 31-nucleotide deletion homologous to the DEN4Δ30 deletion (∆30). Genome-length, capped, RNA transcripts were synthesized from the plasmid p2Δ30-7169 and purified
  Other Names: rDEN2Δ30-7169 Lot DEN2#121A

SUMMARY:
The primary objective is to determine, among dengue-naïve adults in an endemic population, the protective efficacy of TetraVax-DV TV005 vaccine against dengue infection induced by a live recombinant attenuated rDEN2∆30-7169 attenuated virus strain administered 6, 12, or 24 months after vaccination.

Secondary objectives are:

1. Determine the durability of protection of TetraVax-DV TV005.
2. Evaluate the safety of TetraVax-DV TV005 in dengue-naïve volunteers in a dengue endemic population.
3. Evaluate the safety of the rDEN2∆30-7169 attenuated virus strain in a dengue endemic population.

DETAILED DESCRIPTION:
This is a single center, Phase II, placebo-controlled, double-blind study to evaluate the ability of a single dose of TetraVax-DV TV005 vaccine to protect against infection induced by a live recombinant attenuated rDEN2∆30-7169 attenuated virus strain administered 6, 12, and 24 months after vaccination. TetraVax-DV TV005 will contain 103 PFU of rDEN1∆30, 104 PFU of rDEN2/4∆30(ME), 103 PFU of rDEN3∆30/31-7164 and 103 of rDEN4∆30. The dose of rDEN2∆30-7169 attenuated virus strain (DENV-2) will be 103 PFU. The placebo group will receive Plasma-Lyte A Injection pH 7.4.

The study population will be comprised of 192 healthy male and healthy non-pregnant, non-lactating female dengue-naïve adult volunteers aged 18-45 years, inclusive, from dengue-endemic Dhaka, Bangladesh. After providing written informed consent, volunteers will undergo eligibility screening, including medical history, physical examination, hematology testing, liver function testing, hepatitis B and C screening, and serology screening for previous dengue infection. Pregnancy testing will be performed on females with childbearing potential. All screening tests must be performed within 60 days prior to vaccination.

Eligible volunteers will be enrolled to receive TetraVax-DV TV005 or placebo (2:1) on an outpatient basis in one of three cohorts based on intended treatment with the attenuated virus strain timepoint (6, 12 or 24 months). The sequence of treatment assignments to either TV005 or placebo will be generated using block randomization. Randomization will occur sequentially at the time of study enrollment (vaccination) using a pre-generated list. All enrolled volunteers will be followed for 3 years post-vaccination for safety.

At 6, 12, and 24 months post-vaccination, volunteers will be re-screened for treatment with the attenuated virus strain with a live recombinant attenuated DENV-2 virus strain (rDEN2Δ30-7169). Volunteers will receive treatment with the attenuated virus strain in three separate treatment groups each consisting of 33 randomly-selected, eligible vaccine and placebo recipients (2:1) from the three independently vaccinated cohorts. Following treatment with the attenuated virus strain, designated study staff will make home visits to study participants to collect fever and AE information once per day up to day 16. A total of 66 vaccine and 33 placebo recipients (52% of enrolled population) will receive the attenuated virus strain.

Administration of the attenuated virus strain to volunteers at 12 and 24 months is contingent upon DSMB approval following review of all cumulative safety data from those volunteers treated with the attenuated virus strain at 6 months. Volunteers who receive placebo and are subsequently treated with the attenuated virus strain will be offered the TetraVax-DV TV005 vaccination 2 months after their attenuated virus strain dose. All volunteers who receive treatment with the attenuated virus strain will be followed for a minimum of one year post-treatment with the attenuated virus strain for safety (included in the overall 3 years of safety follow up).

Volunteers receiving treatment with the attenuated virus strain will be closely monitored following treatment with the attenuated virus strain and will be admitted to a local hospital for closer observation should they meet admission criteria. Administration of the attenuated virus strain to volunteers at 12 and 24 months is contingent upon DSMB approval following review of all cumulative safety data from those volunteers treated with the attenuated virus strain at 6 months. Volunteers who receive placebo and are subsequently treated with the attenuated virus strain will be offered the TetraVax-DV TV005 vaccination 2 months after their attenuated virus strain dose. All volunteers who receive treatment with the attenuated virus strain will be followed for a minimum of one year post-treatment with the attenuated virus strain for safety (included in the overall 3 years of safety follow up).

ELIGIBILITY:
Inclusion Criteria:

-

All of the following inclusion criteria must be met for a volunteer to be eligible for study participation:

1. Adult male or female between 18 and 45 years of age, inclusive.
2. Good general health as determined by physical examination, laboratory screening, and review of medical history.
3. Available for the duration of the study and willing to consent to a potential inpatient admission following receipt of the attenuated virus strain.
4. Willing to participate in the study as evidenced by signing the informed consent document.
5. Females of childbearing potential only: Willing to use effective contraception for at least 30 days prior to and 28 days following receipt of the investigational product.

Exclusion Criteria:

-

A volunteer will not be eligible for study participation if any of the following criteria are met:

1. Serologic evidence of previous wild-type dengue.
2. Females Only: Currently lactating, breastfeeding or pregnant, as determined by positive urine human choriogonadotropin (CG) test.
3. Positive test result on rapid point-of-care NS1 dengue test performed on study day 0.
4. Interim history of fever without a known cause since screening visit.
5. Evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, rheumatologic, autoimmune, or renal disease by history, physical examination, and/or laboratory studies.
6. Behavioral, cognitive, or psychiatric disease that in the opinion of the investigator affects the ability of the subject to understand and cooperate with the requirements of the study protocol.
7. Screening laboratory values of Grade 1 or above for absolute neutrophil count (ANC), ALT, or platelets as defined in this protocol.
8. Any other condition that in the opinion of the investigator would jeopardize the safety or rights of a volunteer participating in the trial or would render them unable to comply with the protocol.
9. Any significant alcohol or drug abuse in the past 12 months which has caused medical, occupational, or family problems, as indicated by subject history.
10. History of a severe allergic reaction or anaphylaxis.
11. Hepatitis C virus (HCV) infection, by screening and confirmatory assays
12. Hepatitis B virus (HBV) infection, by Hepatitis B surface antigen (HBsAg) screening.
13. Self-reported or suspected immunodeficiency, or receipt of immunosuppressive therapy within the preceding 6 months, or long-term systemic corticosteroid therapy.
14. Current use of anticoagulant medications.
15. Use of aspirin and/or non-steroidal anti-inflammatory medications within 7 days of vaccination or anticipated receipt within 14 days following vaccination.
16. Receipt of a live vaccine within 28 days or a killed vaccine within the 14 days prior to vaccination or anticipated receipt of any vaccine during the 28 days following vaccination.
17. Previous receipt of a licensed or experimental dengue vaccine.
18. Asplenia.
19. Receipt of blood products, including transfusions or immunoglobulin within 90 days prior to receipt of investigational product or anticipated receipt during the study period.
20. Anticipated receipt of any investigational agent in the 28 days before or after receipt of investigational product.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 192 (Actual)
Dates: Start 2021-12-11 (Actual); Primary Completion 2023-11-20 (Actual); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Frequency of viremia | 28 days following challenge.
  Proportion of volunteers with viremia following treatment with the attenuated virus strain among those who received TV005 versus placebo at vaccination. Viremia will be measured by qRT-PCR.

SECONDARY OUTCOMES:
Quantity of Viremia | 28 days following challenge
  Quantity of viremia following treatment with the attenuated virus strain. Quantity of viremia will be measured by qRT-PCR.
Duration of viremia | 28 days following challenge
  Number of days viremic following treatment with the attenuated virus strain.
Frequency of volunteers with adverse events | 28-days post receipt of TV005 or placebo
  Proportion of volunteers in each arm experiencing adverse events.
Frequency of volunteers with adverse events | 28-days post receipt of challenge
  Proportion of volunteers in each arm experiencing adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Beth Kirkpatrick, MD, Principal Investigator — University of Vermont; Rashidul Haque, MD, Principal Investigator — International Centre for Diarrhoeal Disease Research
Locations (1):
- Icddr,B, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No